CLINICAL TRIAL: NCT04658654
Title: A Proof of Concept Phase II Study With the PDE4 Inhibitor Roflumilast in Patients With (Amnestic) Mild Cognitive Impairment (MCI) or Mild Dementia
Brief Title: Cognitive Effects of Roflumilast in (a)MCI and Mild Dementia Patients
Acronym: ROMEMA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 72476
Record Dates: First submitted 2020-08-31; First posted 2020-12-08 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Mild Cognitive Impairment; Mild Dementia; Amnestic Mild Cognitive Disorder
Keywords: MCI, amnestic MCI, mild dementia
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Roflumilast; Phosphodiesterase 4 Inhibitors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo oral capsule, once daily for 24 weeks
  Interventions: Drug: Placebo oral tablet
- Roflumilast 50ug (Experimental): Roflumilast (50 microgram) oral capsule, once daily for 24 weeks
  Interventions: Drug: Roflumilast
- Roflumilast 100ug (Experimental): Roflumilast (100 microgram) oral capsule, once daily for 24 weeks
  Interventions: Drug: Roflumilast

INTERVENTIONS:
Drug: Roflumilast — chronic intervention (24 weeks): roflumilast capsule
  Other Names: EU: Daxas; US: Daliresp; PDE4 inhibitor
  Arms: Roflumilast 100ug; Roflumilast 50ug
Drug: Placebo oral tablet — Pill with inactive ingredients to mimic same appearance of roflumilast capsule
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The aim of the current project is to validate whether chronic intake (24 weeks) roflumilast (PDE4 inhibitor) can improve cognition in patients with (amnestic) mild cognitive impairment (MCI) and in patients with mild dementia. The project will demonstrate whether episodic memory, but also attention, information processing or executive function improves with chronic administration of roflumilast in (a)MCI and mild dementia patients.

ELIGIBILITY:
Inclusion Criteria:

* 50 to 90 years of age
* Willingness (including the informal caregiver) to sign an informed consent
* Body mass index (BMI) between 18.5 and 35
* MMSE of 20 or higher
* Clinical (amnestic)MCI or mild dementia diagnosis
* Memory performance on the delayed recall in the clinically relevant 15 words VLT of 1 or more SD below the average
* Clinical dementia rating (CDR) scale total score of 0.5 or 1
* Fazekas of 2 or lower

Exclusion Criteria:

* Normal Pressure Hydrocephalus (NPH)
* Fazekas of 3 or higher
* Morbus Huntington
* Parkinson's disease
* HIV/AIDS
* Hepatitis C & B
* Recent Transient Ischemic Attack (TIA) (< 2 years)
* Cerebrovascular Accident (CVA) (< 2 years)
* TIA/CVA followed by cognitive decline (within 3 months)
* Chronic Obstructive Pulmonary Disease (COPD) gold criteria 3 or 4 and severe asthma
* History of schizophrenia, bipolar disorder or psychotic symptoms not otherwise specified or previous treatment for these diseases (lifetime)
* Current radiotherapy
* Current affective disorder (i.e. anxiety or major depression)
* Cognitive problems due to alcohol abuse, brain tumor, epilepsy, encephalitis or lack of capacity to consent to participation.
* Current treatment with (or illicit use of) cannabis, opiates, benzodiazepines, MDMA and cocaine
* Patients with moderate or major liver impairments will be excluded (e.g. Child-Pugh B and C).
* Use of medication showing strong inhibition of either CYP3A4 or CYP1A2
* Patients with rare hereditary problems of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
* Patients participating in other drug studies
* If patient does not have the possibility to be accompanied by the same informal caregiver during all test days

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2021-11-19 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Verbal Learning Test (VLT) (15 words) | Change from baseline to 24 weeks of chronic intake

SECONDARY OUTCOMES:
Alzheimer's disease Assessment Scale- Cognitive Sub-scale (ADAS-Cog scale) | Change from baseline to 24 weeks of chronic intake
Mini Mental State Examination (MMSE) | Change from baseline to 24 weeks of chronic intake
Pattern Separation Task | Change from baseline to 24 weeks of chronic intake
Trail-Making Test (TMT) | Change from baseline to 24 weeks of chronic intake
Letter Digit Substitution Test (LDST) | Change from baseline to 24 weeks of chronic intake
Hospital Anxiety and Depression Scale (HADS) | Change from baseline to 24 weeks of chronic intake
Alzheimer's disease co-operative study activities of daily living (ADCS-ADL) scale | Change from baseline to 24 weeks of chronic intake
Neuropsychiatric Inventory (NPI) | Change from baseline to 24 weeks of chronic intake
QoL-AD | Change from baseline to 24 weeks of chronic intake
EuroQol | Change from baseline to 24 weeks of chronic intake
Boston Naming Task | Change from baseline to 24 weeks of chronic intake

OTHER OUTCOMES:
Conversion to Alzheimer's disease (AD) | 24 weeks
Pharmacokinetic validation of roflumilast and its active metabolite roflumilast N-Oxide in plasma | Acute, 12 weeks chronic intake and 24 weeks chronic intake
Tau in tears | Change from baseline to 24 weeks of chronic intake

CONTACTS AND LOCATIONS:
Overall Officials: Inez Ramakers, Dr., Principal Investigator — Psychiatry and Neuropsychology, FHML, Maastricht University, the Netherlands.; Frans Verhey, Prof. Dr., Study Director — Psychiatry and Neuropsychology, FHML, Maastricht University, the Netherlands; Arjan Blokland, Prof. Dr., Principal Investigator — Neuropsychology & Psychopharmacology, FPN, Maastricht University, The Netherlands; Jos Prickaerts, Prof. Dr., Principal Investigator — Psychiatry and Neuropsychology, FHML, Maastricht University, the Netherlands.
Locations (1):
- University of Maastricht, Faculty of Psychology and Neuropsychology, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Possemis N, Verhey F, Prickaerts J, Blokland A, Ramakers I. A proof of concept phase II study with the PDE-4 inhibitor roflumilast in patients with mild cognitive impairment or mild Alzheimer's disease dementia (ROMEMA): study protocol of a double-blind, randomized, placebo-controlled, between-subjects trial. Trials. 2024 Mar 4;25(1):162. doi: 10.1186/s13063-024-08001-3. PMID 38438923